CLINICAL TRIAL: NCT02759692
Title: Clinical Evaluation of Two Approved Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5829
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Test/Control/Test) (Active Comparator): Subjects randomly assigned to the TEST Contact Lens or the CONTROL Contact Lens in the TEST / CONTROL / TEST wearing sequence will wear lenses as daily disposable on both eyes for approximately one week each with no washout period between lenses for at least five days, and 8 hours per day.
  Interventions: Device: TEST Contact Lens; Device: CONTROL Contact Lens
- Group 2 (Control/Test/Control) (Active Comparator): Subjects randomly assigned to the TEST Contact Lens or the CONTROL Contact Lens in the CONTROL / TEST / CONTROL wearing sequence will wear lenses as daily disposable on both eyes for approximately one week each with no washout period between lenses for at least five days, and 8 hours per day.
  Interventions: Device: TEST Contact Lens; Device: CONTROL Contact Lens

INTERVENTIONS:
Device: TEST Contact Lens
  Other Names: senofilcon A
Device: CONTROL Contact Lens
  Other Names: stenfilcon A

SUMMARY:
Adaptive, randomized, subject-masked, dispensing study to evaluate the short-term, clinical performance of two FDA-approved contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between (and including) 18 and 39 years of age.
4. The subject must be an adapted wearer of spherical soft contact lenses in both eyes. That is, the subject must wear their habitual lenses at least five (5) days per week and eight (8) hours per day, worn for at least 30 days immediately preceding the study.
5. Have vertex-corrected distance refraction that allows a plano over-refraction with the available contact lens powers of -1.00 to -6.00 Diopters (D) in each eye.
6. Have refractive astigmatism, if present, of less than or equal to 1.00 D in each eye.
7. The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or breastfeeding (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any autoimmune disease or use of medication, which may interfere with contact lens wear.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or aphakia.
5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.).
6. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
7. Any ocular infection.
8. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
9. Monovision, multi-focal, toric, or extended wear contact lens correction.
10. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
11. History of binocular vision abnormality or strabismus that is likely to affect successful contact lens wear.
12. Any infectious disease (e.g., hepatitis, tuberculosis) or contagious immunosuppressive diseases (e.g., HIV) by self-report.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 283 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Becky Bizzle, OD, Montgomery, Alabama
  - Complete Family Eye Care of Fruit Cove, Jacksonville, Florida
  - Golden Family Eyecare, Sarasota, Florida
  - St. Lucy's Vision Center, Tampa, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - VisualEyes, Inc., Roswell, Georgia
  - Advantage Eyecare Associates, LLC, Neodesha, Kansas
  - Sacco Eye Group, Vestal, New York
  - Advanced Family Eye Care, Denver, North Carolina
  - Total Eye Care PA, Memphis, Tennessee
  - Brian Frazier, OD, Jacksonville, Texas
  - Timothy R. Poling, OD, Salem, Virginia
  - Ziegler Leffingwell Eyecare, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 283 subjects were enrolled into this study. Of the enrolled subjects all were dispensed at least one study lens. Of the dispensed subjects 276 subjects completed the study and 7 subjects were discontinued.
Groups:
- Senofilcon A/ Stenfilcon A/ Senofilcon A: Subjects randomized to this sequence received the senofilcon A lens during the first period, the stenfilcon A lens during the second period and the senofilcon A lens during the third period.
- Stenfilcon A/ Senofilcon A/ Stenfilcon A: subjects randomized to this sequence received the stenfilcon A lens during the first period, the senofilcon A lens during the second period and the stenfilcon A lens during the third period.
Period: Period 1
Arm/Group | Senofilcon A/ Stenfilcon A/ Senofilcon A | Stenfilcon A/ Senofilcon A/ Stenfilcon A
Started | 141 | 142
Completed | 138 | 140
Not Completed | 3 | 2
Not completed — Test article no longer available | 1 | 1
Not completed — No longer meets eligibility criteria. | 1 | 0
Not completed — Miss-Randomized | 1 | 1
Period: Period 2
Arm/Group | Senofilcon A/ Stenfilcon A/ Senofilcon A | Stenfilcon A/ Senofilcon A/ Stenfilcon A
Started | 138 | 140
Completed | 137 | 139
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Test article no longer available | 0 | 1
Period: Period 3
Arm/Group | Senofilcon A/ Stenfilcon A/ Senofilcon A | Stenfilcon A/ Senofilcon A/ Stenfilcon A
Started | 137 | 139
Completed | 137 | 139
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184
  Male | 92
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Black or African American | 30
  White | 237
Region of Enrollment [Number; unit: Participants]
  United States | 276

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. Please note this was a 2 treatment by 3 period study design. Therefore, some subjects were randomized to receive one of the study lenses twice, hence the number of observations were summarized per lens type. For the senofilcon A lens 132+136+132=400 (Observations- 1 per subject per period) from period 1, 2 and 3 respectively. For the stenfilcon A lens 136+132+136=404 (observations) from period 1, 2 and 3 respectively.
Time Frame: 7-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Observations
Groups:
- Senofilcon A: Subjects that received the senofilcon A lens during any of the three study periods.
- Stenfilcon A: Subjects that received the stenfilcon A lens during any three of the study periods.
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 132 | 136
Number analyzed (Observations) | 400 | 404
Units on a Scale | 72.5 (27.9) | 63.8 (30.1)

2. Primary Outcome: Overall Quality of Vision
Description: Overall quality of vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. Please note this was a 2 treatment by 3 period study design. Therefore, some subjects were randomized to receive one of the study lenses twice, hence the number of observations were summarized per lens type. For the senofilcon A lens 132+136+132=400 (Observations- 1 per subject per period) from period 1, 2 and 3 respectively. For the stenfilcon A lens 136+132+136=404 (observations) from period 1, 2 and 3 respectively.
Time Frame: 7-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Observations
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 132 | 136
Number analyzed (Observations) | 400 | 404
Units on a Scale | 67.5 (20.6) | 62.1 (22.3)

3. Secondary Outcome: Individual Patient Reported Outcomes (Items 1-5)
Description: Individual patient reported outcomes questions were used to assess patient-experience attributes of soft contact lenses (e.g. comfort and vision). Items were assessed at the 7-Day follow-up using a 5-point scale of either (1) Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree or (2) Poor, Fair, Good, Very Well, Excellent. Subject's responses for each item were dichotomoized into top-two-box (T2B) response where T2B=1 if a subject responded positively to the question which is dependent on the response set) and T2B=0 otherwise. The percentage of T2B for each item and lens was reported. The following items were asked: ([] indicate the question was abbreviated due to space)1."These Lenses Were Very Comfortable At The End Of The Day" 2."The Comfort of these lenses decreased throughout the day" 3. The lenses were very comfortable from the time I got up to the time I went to bed" 4. "Overall Comfort" 5. "Comfort throughout the Day"
Time Frame: 7-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Responses
Units Other Than Participants: Observations
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 132 | 136
Number analyzed (Observations) | 400 | 404
Percentage of Responses
  [Lenses were very comfortable at end of day] | 75.1 | 65.1
  [Comfort of lenses decreased during day] | 68.5 | 58.1
  [Comfortable lenses when i got up to bed time] | 75 | 61.1
  Overall Comfort | 79.5 | 67.5
  Comfort Throughout the Day | 72.3 | 58.2

4. Secondary Outcome: Individual Patient Reported Outcomes (Items 6-10)
Description: Individual patient reported outcomes questions were used to assess patient-experience attributes of soft contact lenses (e.g. comfort and vision). Items were assessed at the 7-Day follow-up using a 5-point scale of either (1) Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree or (2) Poor, Fair, Good, Very Well, Excellent. Subject's responses for each item were dichotomoized into top-two-box (T2B) response where T2B=1 if a subject responded positively to the question which is dependent on the response set) and T2B=0 otherwise. The percentage of T2B for each item and lens was reported. The following items were asked: ([] indicate the question was abbreviated due to space)6. "Comfort at the end of the day" 7. They remained comfortable from the moment I put them in until the moment I took them out" 8."Comfort from activity to activity" 9. Comfort across different environments" 10."Comfort while working on a computer"
Time Frame: 7-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Responses
Units Other Than Participants: Observations
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 132 | 136
Number analyzed (Observations) | 400 | 404
Percentage of Responses
  [Remained Comfortable from Insertion to Removal] | 79.3 | 69.8
  Comfort Activity to Activity | 81.6 | 69.8
  Comfort Across Different Environments | 78.3 | 66.9
  [Comfort Working on a computer] | 79.3 | 70.3
  [Satisfied with Distance Visions at Insertion] | 91.3 | 90.2

5. Secondary Outcome: Individual Patient Reported Outcomes (Items 11-14)
Description: Individual patient reported outcomes questions were used to assess patient-experience attributes of soft contact lenses (e.g. comfort and vision). Items were assessed at the 7-Day follow-up using a 5-point scale of either (1) Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree or (2) Poor, Fair, Good, Very Well, Excellent. Subject's responses for each item were dichotomoized into top-two-box (T2B) response where T2B=1 if a subject responded positively to the question which is dependent on the response set) and T2B=0 otherwise. The percentage of T2B for each item and lens was reported. The following items were asked: ([] indicate the question was abbreviated due to space). 11."I was very satisfied with my distance vision when i first put these lenses in my eyes. 12."I was very satisfied by the clarity of my vision at the end of the day" 13."I was satisfied with the quality of my vision at night" 14."With these lenses, I felt very confident to drive at night"
Time Frame: 7-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Responses
Units Other Than Participants: Observations
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 132 | 136
Number analyzed (Observations) | 400 | 404
Percentage of Responses
  [Satisfied with Distance Vision] | 91.3 | 90.2
  [Satisfied with Clarity of Vision at end of day] | 85.8 | 77.3
  [Satisfied with my Quality of Vision at Night] | 89.9 | 84.2
  [Confidence to Drive at Night with these lenses] | 91.3 | 86.9

6. Secondary Outcome: Individual Patient Reported Outcomes (Items 15-17)
Description: Individual patient reported outcomes questions were used to assess patient-experience attributes of soft contact lenses (e.g. comfort and vision). Items were assessed at the 7-Day follow-up using a 5-point scale of either (1) Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree or (2) Poor, Fair, Good, Very Well, Excellent. Subject's responses for each item were dichotomoized into top-two-box (T2B) response where T2B=1 if a subject responded positively to the question which is dependent on the response set) and T2B=0 otherwise. The percentage of T2B for each item and lens was reported. The following items were asked: ([] indicate the question was abbreviated due to space). 15."Clarity of vision during daily activities" 16."Clarity of vision in dim or low lighting conditions" 17. "Clarity of visions when driving at night".
Time Frame: 7-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Responses
Units Other Than Participants: Observations
Arm/Group | Senofilcon A | Stenfilcon A
Number analyzed (Participants) | 132 | 136
Number analyzed (Observations) | 400 | 404
Percentage of Responses
  Clarity of Vision During Daily Activities | 85.6 | 74.5
  [Clarity of Vision in Dim or Low Lighting] | 83.3 | 73.8
  Clarity of Vision When Driving at Night | 81.5 | 70.8

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 30 days per subject.
Arm/Group | Senofilcon A | Stenfilcon A
Serious Adverse Events (participants affected / at risk) | 0/141 | 1/142
Other Adverse Events (participants affected / at risk) | 0/141 | 0/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=141) | Stenfilcon A (N=142)
Hospitalization (General disorders) | 0 (0) | 1 (1) — Subjects was hospitalized for an unknown reason, this event was not related to the study lens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days